CLINICAL TRIAL: NCT04543838
Title: Intraoperative Monitoring and Management Protocol to Reduce Strokes (IMMPRES): Pilot Study
Brief Title: IMMPRES: Intraoperative Monitoring & Management to Reduce Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing, funding
Sponsor: Parthasarathy Thirumala (Other)
Responsible Party: Sponsor-Investigator, Parthasarathy Thirumala, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY20070328
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Disease; Intraoperative Hypertension; Cardiac Surgery; Intraoperative Stroke; Perioperative Hypertension; Acute Perioperative Covert Stroke; Perioperative Complication
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomized prospective single-blind clinical trial
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Control will include standard of care pain management during the postoperative period. Participants in this arm will not receive an Electroencephalogram (EEG) and Somatosensory evoked potentials (SSEP).
  Interventions: Other: Standard of Care BP management
- EEG & SSEP monitoring (Experimental): Intervention will include standard of care pain management during the postoperative period. Participants in this arm will receive an Electroencephalogram (EEG) and Somatosensory evoked potentials (SSEP). EEG will be used to manage blood pressure.
  Interventions: Diagnostic Test: Intervention

INTERVENTIONS:
Diagnostic Test: Intervention — Electroencephalogram (EEG) and Somatosensory evoked potentials (SSEP) intraoperative monitoring
  Arms: EEG & SSEP monitoring
Other: Standard of Care BP management — If blood pressure (BP) control is determined to be necessary, standard of care practices to manage it will be implemented
  Arms: Standard of Care

SUMMARY:
The objective of this study is to prospectively evaluate the therapeutic effectiveness of with blood pressure management using intraoperative neurophysiological monitoring with SSEP and EEG to reduce perioperative stroke. The central hypothesis is that perioperative stroke occurs from emboli in the setting of significant hypoperfusion resulting in ischemia, which leads to infarction. The impact of the proposed research is that, if significant SSEP and EEG changes can be used to identify cerebral perfusion, then timely therapeutic interventions to effectively reduce the impact of perioperative stroke can be directed.

DETAILED DESCRIPTION:
If the patient is eligible, interested, and provides consent, they will complete initial preoperative baseline surveys and assessments. These assessments include: Medical History, Medications, Neurological Exam, NIH stroke Scale, Questionnaire for Verifying Stroke-Free Status (QVSFS), Delirium Screen, Modified Rankin Scale, Barthel Index, Cognitive Assessment: The Montreal Cognitive Assessment (MoCA), Depression Scale, and Quality of Life scale. General history, risk factor profile and physical examination (H&P) will be performed prior to entering the study. Neurological examinations, NIHSS, Modified Rankin Scale and Barthel Index will be performed by study neurologist. A Questionnaire for Verifying Stroke-Free Status (revised Questionnaire for Verifying Stroke-Free Status (QVSFS)), QOL assessment, Delirium and Cognitive assessment will be administered to each potentially eligible patient by a research coordinator. Subjects of child bearing age will complete a pregnancy test.

Baseline surveys and assessments will collected during a pre-operative session, either in conjunction with a pre-op clinic visit in-person prior to surgery during their surgical admission. This will allow maximum flexibility in timing, without interfering with clinical care.

Clinically collected data will be abstracted from the electronic medical record (EMR) for research purposes. We will review the patients preoperative medical records to screen patients for the use of intraoperative monitoring. This is currently a standard clinical practice. After enrollment, the subject will be randomized into the control or intervention group. Subjects will be computer randomized to condition 1:1. It will take approximately a half an hour to complete surveys and study procedures. On the day of surgery, EEG and somatosensory evoked potentials assessments will be performed preoperatively.

Procedure: The cardiac surgeons who will be performing surgery will be informed by the principal investigator. The medical management of patients before, during, and after the procedure will be continued as routine medical care in standard medical therapy group. In the intervention group, standard medical therapy with intraoperative monitoring and management protocol will be done. Our IMMP will be a) intraoperative monitoring with SSEP and EEG during surgery and continued for 4 hours after; b) management protocol will be treating patients based on a SSEP and/or EEG changes. In patients with bilateral SSEP and/or EEG changes, we will aim for a MAP target of the greater of 20% above the patient's preoperative baseline or an absolute threshold of 80 mmHg. In patients with persistent unilateral SSEP and/or EEG changes, the higher MAP target will be maintained followed by immediate post-operative evaluation for stroke.

In the control group, the patient will receive standard of care.

Post-Procedure/Pre-Discharge: Brief history and physical examination daily while patient is in hospital. Neurological examination performed by study Neurologist. Delirium screen will be performed. NIH Stroke Scale (NIHSS) performed by study neurologist 18 to 54 hours post procedure. MRI will be performed before discharge. The MRI will be completed at the MRI Research Center.The Cognitive Assessment: The Montreal Cognitive Assessment (MoCA) will be performed.

Follow-up: At 30 days post-op: Modified Rankin Scale, Barthel Index, Questionnaire for Verifying Stroke-Free Status (QVSFS), Quality of Life Assessment, and Cognitive Assessment: The Montreal Cognitive Assessment (MoCA) will be performed.

Follow-up: At 1 year: Neurological exam, Modified Rankin Scale, Barthel Index, TIA/Stroke Questionnaire, Quality of Life Assessment and cognitive evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Cardiac surgery at UPMC
* Patients who are 18 years of age or older at screening
* Patients with the ability to provide written informed consent

Exclusion Criteria:

* Patient who, as determined by the investigators, are noncompliant or unable to complete follow-up assessments
* Patient with history of dementia or other cognitive impairment. History of dementia will be determined by medical record review.
* Patients who, as determined by the investigators, are unable to complete the preoperative testing
* Have an implanted medical electronic device
* Have indwelling or implanted metal in their body that is not MRI-compatible
* Have claustrophobia. This will be measured by utilizing the standard screening questionnaire for MRI.
* Develop back pain when lying flat for more than 1 hour
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parthasarathy Thirumala, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Started | 0 | 19
Completed | 0 | 0
Not Completed | 0 | 19

BASELINE CHARACTERISTICS:
Population: The data involving EEG & SSEP monitoring was not collected prior to this study's discontinuation
Groups:
- Total: Total of all reporting groups
Arm/Group | EEG & SSEP Monitoring | Standard of Care | Total
Number analyzed (Participants) | 0 | 19 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 19 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 0 | 16 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 19 | 19
Barthel Index [Mean (Standard Deviation); unit: score on scale] — Barthel Index for Activities of Daily Living; range 0-100. 0 indicates total dependency, 100= totally independent (lower number is worse).
  score on scale |  | 97.37 (5.10) | 97.37 (5.10)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a New Clinical Stroke, New Overt Stroke, and Death
Description: Proportion of patients with a new clinical stroke, new overt stroke, and death will be abstracted from subject EMR.
Time Frame: post-operative day 30
Population: Data not collected due to staffing changes; we have no ability to further ability to collect missing data
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Patients With Cognitive Decline
Description: Proportion of patients with cognitive decline will be assessed by observing patients who score up to 2 points or more on the Montreal Cognitive Assessment
Time Frame: post-operative 1 year
Population: 1-year follow up data was not collected due to staffing changes; we have no ability to further ability to collect missing data
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Patients With Transient Ischemic Attack
Description: Proportion of patients with transient ischemic attack will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Patients With Delirium
Description: Proportion of patients with delirium will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: delirium data was not collected due to staffing changes; we have no ability to further ability to collect missing data
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of Patients With Clinical Stroke
Description: Proportion of patients with clinical stroke will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of Patients With Composite of Clinical Stroke
Description: Proportion of patients with composite of clinical stroke will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Proportion of Patients With MACE (Death From Any Cause, Non-fatal MI and Stroke)
Description: Proportion of patients with MACE (death from any cause, non-fatal MI and stroke) will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Proportion of Patients With a Decrease in EuroQol 5-dimension (EQ-5D)
Description: Proportion of patients with a decrease in quality of life will be assessed by the EuroQol 5-dimension (EQ-5D). The EQ-5D questionnaire consists of two parts. The first part contains the EQ-5D descriptive system, comprising of 5 questions regarding mobility, selfcare, usual activities, pain, and depression (scores range from 0 to 1). The second part is a vertical, visual analogue scale with the end-points of "best imaginable health state" and "worst imaginable health state" (scores range from 0 to 100; higher values are better). scores.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Proportion of Patients With a Discrete Diffusion-weighted Imaging (DWI) Lesion
Description: Proportion of patients with a discrete DWI lesion will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Overall Volume of DWI Lesion Burden
Description: Overall volume of DWI lesion burden will be abstracted from subject EMR.
Time Frame: post-operative 1 year
Population: as for outcome 2
Arm/Group | EEG & SSEP Monitoring | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Description: no subjects were enrolled in the EEG & SSEP Monitoring Group
Arm/Group | EEG & SSEP Monitoring | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/19
Other Adverse Events (participants affected / at risk) | 0/0 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT04543838/Prot_003.pdf
  • Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT04543838/SAP_001.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT04543838/ICF_002.pdf